CLINICAL TRIAL: NCT05605704
Title: Efficacy of a Treatment Based on Olive Leaf Extracts in the Control of Diabet
Brief Title: Olive Leaf Extracts in the Control of Diabet
Acronym: Dia-Athr
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, clinical proffesor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Diab-Atherolive
Record Dates: First submitted 2022-09-22; First posted 2022-11-04 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: diabetes; Atherolive
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: In each study population, the patient will be assigned to one of two treatments (atherolive or placebo) using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.
Who Masked: Participant
Masking Description: Active Comparator: atherolive group Placebo Comparator: placebo group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- atherolive (Active Comparator): In this Arm the patient will receive the study drug (atherol) that will be prescribed at a dose of 400 mg, once a day for 3 months.
  Interventions: Drug: Atherolive
- placebo atherolive (Placebo Comparator): In this Arm patients will receive the placebo at a dose of 400 mg once a day for 3 months.
  Interventions: Drug: Placebo Atherolive

INTERVENTIONS:
Drug: Atherolive — The patient will be assigned using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months.
  Arms: atherolive
Drug: Placebo Atherolive — The patient will be assigned using a computer-generated randomization list (1: 1 allocation). The investigator who has the randomization code is not involved in other study procedures and does not interact with participants. The placebo will be prescribed at a dose of 400 mg once a day for 3 months.
  Arms: placebo atherolive

SUMMARY:
This study will be carried out in 2 emergency departments (at the exit of the emergency room) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

Patients over 18 years of age with:

-Diabets

DETAILED DESCRIPTION:
This study will be carried out in 2 emergency departments (at the exit of the emergency room, patients included in the GR2 study) and 2 external consultations (endocrinology of the CHU FB Monastir and diabetology consultation, Jemmal hospital).

All the population will benifit of a biological assessment which include:

* Complete lipid profile, blood sugar, creatinine
* HbA1c (if the patient is diabetic).
* Inflammatory assessment: reactive protein C One population will be rendomized:The population with diabetes. In each study population, the patient will be assigned to one of two treatments (atherolive or placebo). The study drug (atherol) will be prescribed at a dose of 400 mg, once a day for 3 months. The placebo will be prescribed identically.

Continuous blood glucose monitoring to measure indices of glycemic variability is performed at baseline. These patients will be equipped with an iPro continuous glycemic monitoring

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age with:
* diabetes.

Exclusion Criteria:

* Exclusion criteria: None.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-09-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
rate of continuous glycemic monitoring and Hemoglobin A1C | 90 days
  Patients will be fitted with an iPro continuous glycemic monitoring (CGM) recorder (Medtronic, Northridge, CA) for 24 consecutive hours on an outpatient basis . A CGM (Enlite Sensor) sensor is inserted into abdominal (or arm) fatty tissue subcutaneously and calibrated according to Medtronic standard operating guidelines. The iPro Continuous Glucose Recorder measures interstitial subcutaneous tissue glucose levels continuously, recording values every 5 minutes, over a range of 40-400 mg/dL.recorded data will be downloaded for analysis of glucose profile and glucose excursion parameters with the CareLink iPro system. Analysis will be performed on the data obtained within the 24-hour period after placement.

SECONDARY OUTCOMES:
variation in lipid balance | 90 days
  Rate of variation in lipid balance
rate of hospitalization for cardiovascular disease and adverse effects | 90 days
  , rate of hospitalization for cardiovascular disease : acute infarction, hypertension, acute stroke as well as number of adeverse events reported

CONTACTS AND LOCATIONS:
Overall Officials: Nouira Semir, Pr, Principal Investigator — University of Monastir
Locations (1):
- Semir Nouira, Monastir, Monastir Tunisia, Tunisia